CLINICAL TRIAL: NCT02409862
Title: Faces: Choices Study
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Technical issues preventing recruitment.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB201600718 -A; 39-2013 SubStudy (Other: University of Florida)
Record Dates: First submitted 2015-03-12; First posted 2015-04-07 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Socioemotional Aging
Keywords: oxytocin; socioemotional functioning; aging

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin Spray (Experimental): This group will receive the single dose of 24 IU oxytocin, self-administered intranasally (IN). Prior to administration a saliva sampling will be done. Afterwards, they will participate in the Choices Study during EEG and eye tracking recording.
  Interventions: Drug: Oxytocin Spray
- Placebo spray (Placebo Comparator): This group will receive the single dose of 24 IU saline, self-administered intranasally (IN). Prior to administration a saliva sampling will be done. Afterwards, they will participate in the Choices Study during EEG and eye tracking recording.
  Interventions: Drug: Placebo Spray

INTERVENTIONS:
Drug: Oxytocin Spray — This group will receive the single dose of 24 IU oxytocin, self-administered intranasally (IN). Prior to administration a saliva sampling will be done. Afterwards, they will participate in the Choices Study during EEG and eye tracking recording.
  Other Names: synthetic oxytocin
  Arms: Oxytocin Spray
Drug: Placebo Spray — This group will receive the single dose of 24 IU placebo, self-administered intranasally (IN). Prior to administration a saliva sampling will be done. Afterwards, they will participate in the Choices Study during EEG and eye tracking recording.
  Other Names: saline spray
  Arms: Placebo spray

SUMMARY:
The neuropeptide oxytocin (OXT), originally known for its role in inducing uterine contractions has been shown to be involved in many of the social capacities that seem to change with age, such as emotion detection and identification, enhanced social memory, empathy, and trust. Thus, age-related changes in the OXT system may underlie differences between young and older adults in socioemotional functioning. Research on the effects of oxytocin in aging is very scarce; therefore, the purpose of this research project is to determine the effects of oxytocin on socioemotional aging. The aim of this research is to examine the behavioral and neural effects of OXT on decisions of trust in social interactions, perceptions of facial trustworthiness, the ability to read faces, and levels of empathy with other people in samples of young and older adults.

DETAILED DESCRIPTION:
Overview: This study has three parts: An initial screening visit and two study visits. All visits to be conducted at the Institute on Aging at the University of Florida.

Screening Visit - Screening: Together with the information obtained in the phone screening, the main purpose of the screening visit is to find out if the participants are eligible to participate in the study.

* One of the investigators trained researchers will ask the participant questions about their health condition, and recent activities.
* The participant will be given instructions and assistance in the collection of saliva to determine the baseline level of cortisol in their body.
* A trained researcher will then ask the participant questions about their personality and experiences in close relationships.
* The participant will then be asked to provide the second saliva sample to find out how the activity of their genes may impact their cognition and behavior during the tasks they engage in as part of the study.
* The researcher will then conduct two cognitive tests (Digit Substitution Task, Verbal Learning Test).
* This will be followed by a blood test to screen for medical conditions that may indicate that the participant should not participate in the study, such as certain blood levels elevated out of normal range. The blood test will also be used to determine the level of oxytocin, testosterone, and estrogen in the participant's body that occur normally.
* The participant will then have a brief consultation with a licensed physician, to go over their medical review. This will not be a clinical doctor visit for routine medical care, but a visit to confirm the participant's healthy medical status to participate in the research study.

Study Visits -

* A researcher will ask the participant to answer a short questionnaire comprising questions about activities and events during the last 24 hours.
* A researcher will ask for the participant to respond to a short questionnaire related to their current mood.
* The participant will be asked to provide a first saliva sample to determine the baseline level of oxytocin in their body on the day of testing.
* The participant will be asked to self-administer either the oxytocin or a placebo, into their nose by using a nasal spray bottle. Oxytocin is a hormone that naturally occurs in the body and has been shown to be relevant for many behaviors, especially in social situations. The participant will be assigned by chance, much like the flip of a coin, to receive either the oxytocin or the placebo during the first study visit. The participant will then receive the other during the second study visit respectively.
* The participant will then be asked to participate in an electroencephalography (EEG) recording session, that is recording of electrical activity along their scalp. An EEG cap, selected for the participant's head size, will be placed on their head. During this part of the study, the participant will sit in a comfortable chair while working on the Choice Task on the computer screen or resting.
* While recording EEG, the participant's eye movements will be monitored with an eye tracker. The eye-tracking camera will be placed so that it can capture the participant's eyes and after a brief calibration procedure will track the participant's eye movements while working on the task or resting.
* The Choice Task will involve making decisions that involve the participant as well as a fellow player. Before the task starts, the participant will receive detailed information and have a chance to ask any questions that they may have about the task or about the EEG and eye tracking procedures. They will also have the chance to work on some practice trials.
* Next, the participant will be asked to provide a second saliva sample to determine the level of oxytocin in their body after they have received the oxytocin or placebo and some time has passed.
* After the Choice Task, the participant will complete a few more questionnaires, including questions about feelings and thoughts about themselves and others, and questions about how they completed the Choice Task and whether they experienced any drug side effects or any discomfort during the EEG or eye tracking.
* The second study visit will take place about a week after the first study visit, and will be identical in procedure.
* Both visits will be followed up by a brief phone call from a researcher about 3 days after the study visit.
* Upon completion of the study, the participant will receive study reimbursement. A researcher will tell the participant about the general goals of the study and answer any questions that they may have.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-33 (for the younger adults) and 60-85 (for the older adults)
* Male
* Caucasian
* English fluency

Exclusion Criteria:

* Severe claustrophobia
* Currently on vasoconstrictors, pseudoephedrine or antidiuretic medication
* Surgery on the brain or any prior serious brain damage or disease
* Dementia or severe cognitive disorders
* History of hyponatremia, Syndrome of Inappropriate Antidiuretic Hormone, psychogenic polydipsia, or motion disorder

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
The change in choices task between baseline and at week 2 | Change between baseline and at week 2
  Interactive computer task that determines willingness to give money to a fellow player.

SECONDARY OUTCOMES:
The change in General Trust Measure Questionnaire between baseline and at week 2 | Change between baseline and at week 2
  Participants will work on the 11-item General Trust Measure (General Trust Measure; Rothstein, 2011), which assesses participants' level of trust on a scale ranging from 1 = strongly disagree to 7 = strongly agree. With a total overall score of 77 being the best possible score, and 11 is the worst overall score.
The change in Empathy Quotient Questionnaire between baseline and at week 2 | Change between baseline and at week 2
  Participants will fill out a 22-item version of the Empathy Quotient (EQ-Short; Wakabayashi et al., 2006), on a scale ranging from 1 = strongly disagree to 5 = strongly agree. With a total overall score of 110 being the best possible score, and 22 is the worst overall score. This measure assesses empathy, as the drive to identify emotions and thoughts in others and to respond to these with an appropriate emotion.
The change in Trait Meta-Mood Scale Questionnaire between baseline and at week 2 | Change between baseline and at week 2
  Participants will respond to seven items from two subscales (Attention to feelings; Clarity of feelings) of the Trait Meta-Mood Scale (TMMS; Salovey, Mayer, Goldman, Turvey, & Palfai, 1995), as a measure of emotional attention and clarity, using a scale ranging from 1 = strongly disagree to 5 = strongly agree. With a total overall score of 35 being the best possible score, and 7 is the worst overall score.
The change in Inclusion of Community in the Self Scale Questionnaire between baseline and at week 2 | Change between baseline and at week 2
  Participants will respond to a modified version of the Inclusion of Community in the Self Scale (#14-ICS; Mashek, Cannaday, & Tangney, 2007). This measure assesses the connectedness an individual feels to other people. Participants will be presented pictures of two circles with different degrees of overlap (representing different extents of connectedness) and will be told that one circle represents themselves and the other circle represents people of a particular age group (young, older). Participants will be asked to mark the picture that best describes their connectedness with the age group specified. This will be repeated for each of the two age groups, counterbalanced across participants. Participants will select a maximum of one picture per age group.
Gift basket task | Week 2
  Participants are given the choice to give their fellow players either a candy or fruit basket.
Donation task | Week 2
  Participants are given the option to donate their reimbursement to a charity.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie C Ebner, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States